CLINICAL TRIAL: NCT01715116
Title: ENHANCED Device Programming to Reduce Therapies and Improve Quality of Life in Implantable Cardioverter Defibrillator Patients: A Prospective, Single-arm Safety Monitoring Study (ENHANCED-ICD Study)
Brief Title: ENHANCED Device Programming to Reduce Therapies and Improve Quality of Life in Implantable Cardioverter Defibrillator (ICD) Patients
Acronym: ENHANCED-ICD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: M. Meine (Other)
Collaborators: Medtronic (Industry); Tilburg University (Other); Julius Center (Other)
Responsible Party: Sponsor-Investigator, M. Meine, Mathias Meine, MD, PhD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12/301
Record Dates: First submitted 2012-10-10; First posted 2012-10-26 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Cardiac Arrhythmias
Keywords: Cardiac arrhythmias; Implantable Cardioverter-Defibrillator; Patient Safety; Quality of life
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enhanced ICD programming (Experimental)
  Interventions: Device: Enhanced ICD programming

INTERVENTIONS:
Device: Enhanced ICD programming — * VT monitor: > 166/min
  * fVT: > 182/min; via VF 60/80 intervals (number of intervals to start ATP after approximately 20 s); 3 x ATP (8 stimuli, 88%, scan 20 ms); shock 1-5: 35 J; redetection 30/40 intervals.
  * VF: > 250/min; via VF 60/80 intervals (number of intervals to start therapy after approximately 15 s); 1 x ATP (8 stimuli, 88%) during charging; all shocks: 35 J; redetection 30/40 intervals
  * SVT/VT discrimination is turned on, high rate time out is "OFF"
  * SVT/VT discrimination single chamber: stability, wavelet; SVT upper rate limit: 222/min
  * SVT/VT discrimination dual/triple chamber: P/R logic, wavelet; SVT upper rate limit: 222/min
  * T wave-oversensing and lead noise discrimination is turned on in all devices.

SUMMARY:
The purpose of this study is to determine whether Enhanced device programming to reduce therapies (i.e. anti tachycardia pacing (ATP) episodes and shocks (both appropriate and inappropriate)) is safe for patients implanted with an Implantable Cardioverter-Defibrillator (ICD). The secondary objective is to examine the impact of Enhanced programming on (i) ATPs and shocks (both appropriate and inappropriate) and (ii) quality of life and distress.

DETAILED DESCRIPTION:
ICD therapy has become the first-line treatment for the prevention of sudden cardiac death both as primary and secondary prevention due to its proven survival benefits as compared to anti-arrhythmic drugs. However, ICD therapy is associated with a number of complications and shocks that may impair patient quality of life and well being but also influence mortality. Hence, reduction of ICD shocks by means of alternative programming of the device is paramount for improving patient-centered outcomes and mortality.

The ENHANCED-ICD study will be a prospective, single-arm safety monitoring study. All patients will receive Enhanced programming. Furthermore, patients will be asked to complete a set of standardized and validated self-report questionnaires prior to ICD implantation, at 3-, 6-, and 12 months post implantation.

ELIGIBILITY:
Inclusion Criteria:

* a primary or secondary prophylactic indication for ICD therapy according to the current European guidelines
* implanted with a Medtronic ProtectaTM ICD/CRT-D device or any future CE-approved and market-released Medtronic ICD/CRT-D devices with SmartShock technology
* between 18-80 years of age
* speaking and understanding Dutch
* providing written informed consent

Exclusion Criteria:

* a life expectancy less than 1 year
* a history of psychiatric illness other than affective/anxiety disorders
* on the waiting list for heart transplantation
* insufficient knowledge of the Dutch language

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of intervention-related safety events | up to 12 months
  Combined safety endpoint: arrhythmic syncope/hospitalization/death/other serious adverse event.

SECONDARY OUTCOMES:
Number of ATPs/shocks | 2 months post implantation
  ATPs/shocks shall be further classified based on: appropriate/inappropriate; successful/unsuccessful.
Number of ATPs/shocks | 6 months post implantation
  ATPs/shocks shall be further classified based on: appropriate/inappropriate; successful/unsuccessful.
Number of ATPs/shocks | 12 months post implantation
  ATPs/shocks shall be further classified based on: appropriate/inappropriate; successful/unsuccessful.
Quality of life | Baseline
  EuroQol 5D (EQ-5D)and Short Form Health Survey 12 (SF-12)
Quality of life | 3 months post implantation
  EuroQol 5D (EQ-5D)and Short Form Health Survey 12 (SF-12)
Quality of life | 6 months post implantation
  EuroQol 5D (EQ-5D)and Short Form Health Survey 12 (SF-12)
Quality of life | 12 months post implantation
  EuroQol 5D (EQ-5D) and Short Form Health Survey 12 (SF-12)
Distress | Baseline
  Hospital Anxiety and Depression Scale (HADS) and Patient Health Questionnaire (PHQ-9)
Distress | 3 months post implantation
  Hospital Anxiety and Depression Scale (HADS)and Patient Health Questionnaire (PHQ-9)
Distress | 6 months post implantation
  Hospital Anxiety and Depression Scale (HADS)and Patient Health Questionnaire (PHQ-9)
Distress | 12 months post implantation
  Hospital Anxiety and Depression Scale (HADS)and Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Meine, MD, PhD, Principal Investigator — University Medical Center; Susanne Pedersen, PhD, Principal Investigator — Tilburg University
Locations (1):
- University Medical Center, Utrecht, Netherlands

REFERENCES:
- [Derived] Chiu CSL, van Dijkhuizen A, Gerrits W, Cramer MJ, Tuinenburg AE, van der Harst P, Meine M. Reducing Unnecessary Implantable Cardioverter-Defibrillator Therapy With ENHANCED Programming: Long-Term Outcomes of the ENHANCED-ICD Study. J Cardiovasc Electrophysiol. 2025 Nov;36(11):2861-2869. doi: 10.1111/jce.70060. Epub 2025 Aug 18. PMID 40820765
- [Derived] Mastenbroek MH, Pedersen SS, van der Tweel I, Doevendans PA, Meine M. Results of ENHANCED Implantable Cardioverter Defibrillator Programming to Reduce Therapies and Improve Quality of Life (from the ENHANCED-ICD Study). Am J Cardiol. 2016 Feb 15;117(4):596-604. doi: 10.1016/j.amjcard.2015.11.052. Epub 2015 Dec 7. PMID 26732419